Study title:

Prevention of metacarpophalangeal joints structure damage in patients with psoriatic arthritis using secukinumab

NCT03623867

Protocol version 4.0 dated 20 Mar 2020

PI: Lai-Shan Tam1

Co-I: Ling Qin<sup>2</sup>, James Griffith<sup>3</sup>, Lin Shi<sup>1</sup>, Wing-Yin Vivian Hung<sup>2</sup>, Man-Yee Lee<sup>4</sup>

- 1. Department of Medicine & Therapeutics, The Chinese University of Hong Kong;
- 2. Department of Orthopedics & Traumatology, The Chinese University of Hong Kong;
- 3. Department of Imaging & Interventional Radiology, The Chinese University of Hong Kong;
- 4. Department of Medicine & Geriatrics, Tai Po Hospital. Hong Kong.

#### Background:

Psoriatic arthritis (PsA) is a chronic inflammatory joint disease associated with psoriasis. PsA is associated with distinctive clinical features including changes in skin and nails, peripheral arthritis, axial disease, dactylitis and enthesitis. Synovial inflammation in peripheral joints is the most prevalent feature of the disease ranging in severity from mild joint inflammation to disabling peripheral arthritis (1). Within 2 years of diagnosis, radiological erosions were developed in 47% of the patients (2). Without proper monitoring and treatment, it will lead to significant structure damage and loss of physical function, and even arthritis mutilans, which is the most severe destructive form of PsA (3). Prevention of structural damage is one of the primary goals of treating PsA patients to maximise health-related quality of life (4).

Detection of bone erosions in PsA patients is usually achieved by conventional radiographs although the sensitivity is low (5). High-resolution peripheral quantitative CT (HR-pQCT) is a novel technique for detailed bone microstructure analysis with high reproducibility in assessing bony erosions (6). With its high spatial resolution of 130 µm, HR-pQCT exhibited a higher sensitivity in detecting erosion compared with radiograph and magnetic resonance imaging (MRI) (7). Recently, Finzel et al. described an indirect method to assess volume based on measurements of the width and depth of the erosions using HR-pQCT (8). Quantitative measurement of erosion volume can also be achieved (6). Using this method, erosion repair under biological disease-modifying antirheumatic drugs (DMARDs) treatment has been demonstrated in patients with rheumatoid arthritis (RA) (8, 9). Bone apposition at the margin of erosions (osteosclerosis) with the formation of a new cortical lining was associated with a decrease in erosion depth or width, which may indicate either periosteal or endosteal repair processes (8, 9). Valid measurement of erosion volume using HR-pQCT will facilitate the testing of treatments that may help to heal erosion. Decrease in erosion volume and the presence of osteosclerosis on HR-pQCT could be promising markers for erosion healing.

Detection of dactylitis is mainly by clinical assessment currently. With the advancement of ultrasound (US) imaging, it is lately discovered that the dactylitis was related with inflammation of pulley system from a pilot study (data not published). However, there are limited study on the change in inflammation of pulley system by US.

Interleukin 17 (IL-17) is a proinflammatory cytokine which produced by type 17 helper T cells (Th17). It is now considered to be a key cytokine in the pathogenesis of a number of autoimmune disorders in humans including PsA (10). IL-17 was also reported to be associated with the presence of joint erosion (11). Recently, secukinumab, an anti–interleukin-17A monoclonal antibody, was reported to be effective in reducing disease activity and decreased the rate of radiographic joint damage compared with placebo (12). However, whether healing of erosion could occur in PsA has never been evaluated. The US-detected longitudinal changes of dactylitis was not reported too.

On the other hand, osteophytes formation at the entheseal regions of the joints in PsA is distinctive feature compared with RA (13). The formation of osteophytes is tightly regulated by anabolic pathways, which resembles the pathogenesis of new bone formation in ankylosing spondylitis (AS). Tumor necrosis factor (TNF) inhibition was unable to halt the structural progression in AS patients (14-16), it also lacked efficacy in stopping the progression of osteophytes in PsA patients (17). Inhibition of IL-17 by secukinumab was effective in the treatment of both AS (18) and PsA (12). Secukinumab also decreased the rate of radiographic joint damage regarding to erosion and joint space narrowing (12). However, it is unknown if it has any effect in the progression of osteophytes. In an animal model, although over-expression of IL-17 alone failed to induce entheseal and periosteal bone formation, inhibition of IL-17 leaded to significant reduction of such bone formation in an IL-23 overexpression model (19). Moreover, IL-17A accelerates bone formation by stimulating the proliferation and osteoblastic differentiation of mesenchymal progenitor cells after injury (20). It is worth exploring if secukinumab could prevent the progression of osteophytes in PsA patients.

# Aims and hypotheses to be tested:

#### **Hypothesis**

IL-17 inhibition by secukinumab could lead to healing of existing erosion, and prevent progression of osteophytes, and resolution of dactylitis in PsA patients.

#### Aims

The aim of this randomized, double-blind, placebo-controlled study is to evaluate the protective effects of secukinumab on the healing of joint erosion and prevention of progression of osteophytes in PsA patients using HR-pQCT and US.

#### **Objectives**

# **Primary outcome**

Difference in changes in the volume of erosions on metacarpophalangeal joints (MCP) 2-4 measured by HR-pQCT at 24 and 48 weeks between secukinumab and placebo group.

# **Secondary outcomes**

- The percentage of erosions with healing determined using HR-pQCT on MCP 2-4 at 24 and 48 weeks including 1). A decrease in erosion volume of ≥0.4 mm³ from baseline, and 2). The presence of grade 2 osteosclerosis at the margin of erosion.
- 2) Changes in volume and width of erosion using HR-pQCT at 24 and 48 weeks;
- 3) Changes in the height of osteophytes using HR-pQCT at 24 and 48 weeks;
- 4) Marginal osteosclerosis (semi-quantitative and quantitative) using HR-pQCT at 24 and 48 weeks;
- 5) Changes in joint space volume using HR-pQCT at 24 and 48 weeks

# **Exploratory outcomes**

- 1) Changes in US-parameters in dactylitis, enthesitis and synovitis at 24 and 48 weeks
- 2) Changes in van der Heijde-Sharp score on radiograph at 24 and 48 weeks.
- 3) Changes in patients-reported-outcomes (SF-36, Psoriatic Arthritis Impact of Disease (PsAID)) and functional disability (HAQ) at 24 and 48 weeks
- 4) Changes in biomarkers (Pro-C2, C-Col10, COMP, MCP-1, Dkk1 and sclerostin) at 24 and 48 weeks

# Plan of Investigation:

<u>Subjects</u> 120 biologic DMARDs naïve PsA patients attending the outpatient clinic of the Prince of Wales Hospital (PWH), North District Hospital (NDH), Tai Po Hospital (TPH), Queen Elizabeth Hospital (QEH) and Tseung Kwan O Hospital (TKOH) who fulfilled the Classification Criteria for Psoriatic Arthritis (CASPAR), will be recruited. The main inclusion criteria are: 1) ≥18 years old; 2) without severe deformity in MCP joints (MCPJ) which would influence the longitudinal assessment of HR-pQCT; 3) with active disease, which is defined as three or more tender joints and three or more swollen joints, despite previous treatment with nonsteroidal anti-inflammatory drugs, disease-modifying antirheumatic drugs. These 120 patients will be screened for the presence of erosion at the head of MCPJ 2-4 using HR-pQCT. The first 40 patients with erosion will be randomised in a 1:1 ratio to secukinumab (n=20) or placebo (n=20) group. Based on a study using high-resolution CT in 41 PsA patients, 41% of the patients had at least one erosion, and 90% of the erosions were in MCPs (5). The resolution of the high-resolution CT is 0.4 mm, which is almost 5 folds lower than HR-pQCT (82 μm). Therefore, we estimated that over 1/3 of the PsA patients will have at least one erosion in MCPs. Thus, screening 120 patients using HR-pQCT should be adequate to recruit 40 patients with erosions on MCPJ 2-4.

All study procedures will be performed in PWH after recruitment from non-PWH site.

Randomisation will be performed using a computer-generated randomisation list provided by the hospital pharmacist, using a permuted blocks design with block sizes of 4 and 6. Allocation concealment will be ensured by the use of sequentially numbered, opaque, sealed envelopes. Treatment will be masked to patients and investigators.

Exclusion criteria are: 1) limited in ability to perform usual self-care, vocational, and avocational activities; 2) pregnancy; 3) previous therapy with biologic; 4) the presence of active inflammatory diseases other than PsA; 5) active infection in 2 weeks before randomization or a history of ongoing, chronic, or recurrent infections including tuberculosis; 6) history of hepatitis B & C; 7) history of malignant disease within the past 5 years (excluding basal cell carcinoma or actinic keratosis, in-situ cervical cancer, or non-invasive malignant colon polyps); 8) contraindications to secukinumab. The concomitant use of oral glucocorticoids (at a dose of ≤10 mg per day of prednisone or its equivalent) and methotrexate (at a dose of ≤25 mg per week) are permitted, provided that the dose will be stable.

The study will be approved by the Ethics Committee of the Chinese University of Hong Kong. Written informed consent will be obtained from all participants according to the Declaration of Helsinki and ICH-GCP guidelines.

<u>Methods</u> This is a 52-week, randomized, placebo-controlled, double-blind study. PsA patients will be randomised to either secukinumab or placebo group. All patients will be evaluated and treated according to the following protocol.

# Study design

#### **Treatment**

The patients will be randomly assigned to the secukinumab group or placebo group. Patients will be followed-up at weeks 2, 4 and then every 12 weeks until week 52. Patients will receive subcutaneous placebo or secukinumab 150 mg once a week from baseline for 4 weeks, and then once every 4 weeks from week 4 onwards. The study flow is shown in Figure 1. Changes in the baseline treatment, e.g. the dosage of conventional synthetic DMARDs (csDMARDs) including methotrexate, leflunomide, hydroxychloroquine, or sulfasalazine or the addition of a new csDMARD (individually or in combination), as well as changes in the dosage or the addition of steroids or nonsteroidal antiinflammatory drugs were allowed after week 12 if the patient cannot achieve minimal disease activity (MDA) (Table 1) (see appendix 1 for the treatment protocol). For patients who fulfil the criteria for biologic DMARDs (bDMARDs) (Appendix 2) and are willing to be started on bDMARDs, the code will be broken, and they can either pay out of pocket or can apply for the Samaritan Fund for financial assistance, provided they must household-based pass financial assessment (http://www.ha.org.hk/visitor/ha\_visitor\_index.asp?Content\_ID=10048&Lang=ENG&Dimension=100). Patients who have started bDMARDs apart from secukinumab will be excluded from the efficacy assessment. Adverse effects will be recorded.

**Evaluation of disease activity and severity** 

At baseline and at each visit, we will quantify the extent of disease by evaluation of the multiple clinical domains of PsA. The following domains will be assessed: pain, physicians' and patients' global assessments, number of tender and swollen joints (using the 68 tender/66 swollen joint count), number of joints irreversibly damaged (baseline and week 52 visit only); enthesitis ((Maastricht Ankylosing Spondylitis Enthesitis Score (MASES), The Leeds Enthesitis Index (LEI) and the Spondyloarthritis Research Consortium of Canada Enthesitis Index (SPARCC Enthesitis Index). ); number of digits with dactylitis; levels of acute phase reactant including erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP) levels, Bath ankylosing spondylitis disease activity index (BASDAI), Bath Ankylosing Spondylitis Functional Index (BASFI) and the modified health assessment questionnaire (M-HAQ. For the skin domain, Psoriasis Area (BSA) and Psoriasis Activity and Severity Index (PASI) will be assessed in baseline and each visit. Quality of life will be assessed at baseline, week 24 and 48 which include HRQoL using the Short Form 36 (SF-36) Health Survey and the Psoriatic Arthritis Impact of Disease (PsAID) [21]. MDA will be used for assessment of treatment efficacy endpoint. A qualified dermatologist will be responsible for performing assessment of skin involvement (BSA, PASI) of the patients.

Composite disease activity will be assessed at baseline and at each visit according to the PASDAS (Table 2) (21). The PASDAS is calculated using the following variables: patient global VAS (0-100), physician global VAS (0-100), 66 swollen joint count, 68 tender joint count, CRP level (mg/ litre), Leeds enthesitis count (0-6), tender dactylitis count (0-20), and the physical component summary (PCS) scale of the Short Form 36 (SF-36) health survey. The PASDAS is then calculated by the formula [22]:

```
PASDAS = (0.18 \times \sqrt{\text{physician global VAS}})
```

```
+ (0.159 × \sqrt{} patient global VAS)

- 0.253 × \sqrt{} SF-36 - PCS) + (0.101

× LN [swollen joint count + 1])

+ 0.048 × LN [tender joint count + 1])

+ (0.23 × LN [Leeds Enthesitis Count + 1])

+ (0.377 × LN [dactylitis count + 1])
```

The PASDAS was developed by GRAPPA based on real patient data from the GRAppa Composite Exercise (GRACE) project and it has been utilised by recent studies to monitor treatment response of biologic DMARDs including secukinumab and golimumab [23, 24].

+  $(0.102 \times LN [CRP + 1] + 2 \times 1.5$ , where LN is the natural logarithm.

At baseline, 24 and 48 weeks, Muscle-skeletal US will be examined for enthesitis, dactylitis and synovitis assessment; while X-rays of the hands, wrists, feet, hip and (X-ray pelvis for those with axial involvement) will be performed for the evaluation of erosion.

# **Laboratory assessments and inflammatory markers**

Laboratory assessments at baseline, 24 and 48 weeks the end of study include fasting blood glucose, fasting lipid profile (total cholesterol, low-density lipoprotein-cholesterol [LDL-C], high-density

lipoprotein-cholesterol [HDL-C], triglycerides), fibrinogen, and uric acid. Total cholesterol is measured by an autoanalyzer enzymatic method. HDL-C is determined enzymatically with polyethylene glycol—modified enzymes. LDL-C is calculated by the Friedewald formula. If the triglyceride levels exceed 4.0mmoles/liter, the LDL levels are measured directly by ultracentrifugal single spin analysis. A total of 16 ml research blood will be collected for the following research use.

It has been suggested that chronic skin inflammation could lead to bone loss by IL-17-mediated inhibition of the WNT signalling pathway [25]. In order to investigate the effects of Secukinumab on the proposed pathway, the levels of WNT-inhibitors including Dickkopf-1 (Dkk1) and sclerostin will be measured with enzyme-linked immunosorbent assays (ELISA).

As joint space narrowing will be assessed (see below), relevant markers of cartilage formation, metabolism and turnover (Pro-C2, C-Col10, COMP and MCP-1) will be measured using ELISA according to the manufacturer's instructions [26, 27].

# Safety Data Collection and Reporting

All possible side effect of the biologic and synthetic DMARDs used the study will be explained to the participants by the research nurse and the treating physician. To monitor the possible side effect, complete blood count, liver function tests and renal function tests will be performed every visit. Chest X-rays will be obtained at baseline and at the end of the study. The treating physician records all nonserious and serious adverse events, all reports of drug exposure during pregnancy, and all reports of misuse and abuse of the Novartis drug, other medication errors and uses outside of what is foreseen in the protocol, if necessary, make treatment adjustments in accordance with the protocol. Serious adverse events are defined as any adverse reaction resulting in any of the following outcomes: a lifethreatening condition or death, a significant or permanent disability, a medically significant event, hospitalization or prolongation of hospitalization, a congenital abnormality, or a birth defect. All adverse events from this trial will be reported to local IRB and Health Authority by the investigator according per requirement as holder of certificate of clinical trial. Any SAEs, reports of drug exposure during pregnancy and reports of Study Drug misuse or abuse, including initial and follow up reports, arising from the Study in subjects exposed to the Study Drug, as soon as it becomes available, but in any event within fifteen (15) calendar days of becoming aware of such information, will be forwarded to Novartis by transmitting it to Novartis Patient Safety team.

# **Erosion assessment by HR-pQCT**

Image acquisition

Metacarpal bone erosion will be assessed at MCP 2-4 of the more severely affected or the dominant hand if both hands are equally affected using a HR-pQCT system (XtremeCT II; Scanco Medical AG, Bruttisellen, Switzerland). This system enables the simultaneous acquisition of CT slices with an isotropic resolution (voxel size) of 82  $\mu$ m. HR-pQCT scanning will be performed by a single investigator who is blinded to all the clinical information of the patients. A single examination will be performed for

measurements of MCP 2-4. An anteroposterior scout view will be used to define the region of interest (ROI). The scan region will be 80 slices distal and 242 slices proximal of the upper margin of the head of MCP3. Scan time will be around 8 min per patient and scan (8). The scans will be performed at baseline, 24 and 48 weeks.

#### Erosion identification and measurement of the width and depth

Erosions are defined as sharply marginated bone lesions with juxta-articular localisation with a cortical break seen in at least two adjacent slices, which are often accompanied by loss of the adjacent trabecular bone. Erosions will be differentiated from physiological breaks indicating entry of blood vessels by the linear shape and occurrence on predilection sites. Pseudo-erosions, structures similar to cortical breaks presented by osteophytes, will be excluded (22). Each of the erosions will be documented at baseline and 48 weeks. Assessment includes the palmar, ulnar, dorsal as well as the radial sides of MCP 2-4 heads investigating overall 322 2D HR-pQCT slices in the transversal, sagittal and coronal plane. Every erosion of each patient will be characterised by the maximal width and depth of the lesion in the axial, sagittal and coronal using the open source DICOM viewer Osirix V3.2 (Rosslyn, VA, USA).

#### Erosion volume

The volume of the erosions will be calculated according to the methodology published by Fouque-Aubert et al (6). The volume of erosions (using the entire volume of interest) will be determined by manually defining the ROI including the erosion (V1) or excluding it (V2). The volume of erosions will be then calculated as: Verosion= V1-V2; V =sum(A\_i\*0.082), where A1\_i or A2\_i is the area on slice i (mm²), including or excluding erosion, and 0.082 mm is the thickness of slice (Figure 2).

#### Osteosclerosis

The signs of bone apposition at the margin of the erosion will be documented (8, 9). Semi-quantitative scoring (0-2 scale) of osteosclerosis will be performed using coronal reconstructions as follows: grade 0 = 0%, grade 1 = 1-75%, grade 2 = 75-100% bone apposition along the surrounding bone (typical images were shown in Figure 3) (23). Quantitative osteosclerosis will also be calculated by choosing the area (width =15 vexols) around bone erosion in MCP2-4 as ROI (24). The density of the ROI will be calculated as the mean pixel attenuation of that area. 3D registration will be applied to obtain a consistent segmentation of the periosteal surface in the vicinity of the cortical break, which is highly important for accurate quantification of bone damage.

# Defining the healing of erosion

This is the first study assessing erosion healing using HR-pQCT. Erosion healing is evidenced by a decrease in erosion volume and the presence of bone apposition at the margin of the erosion. Based on our preliminary data, the smallest detectable change of erosion volume, which was calculated on

the basis of 29 individual erosions as suggested by Bruynesteyn et al. (25), was 0.4 mm<sup>3</sup>. Meanwhile, a grade 2 osteosclerosis means dramatic bone apposition at the erosion margin (>75%). Therefore, a decrease in erosion volume of ≥0.4 mm<sup>3</sup> from baseline, and the presence of grade 2 osteosclerosis at the surface of erosion at 24 or 48 weeks is considered as strong evidence of erosion healing.

#### **Osteophytes**

The maximal height of each osteophyte will be documented by assessing the maximal distance between the surface of the osteophyte and the original cortical bone surface using the open source DICOM viewer Osirix V3.2 (Rosslyn, VA, USA) (17). The change of the maximal height between baseline and 52 weeks will be calculated.

Images will be evaluated by two independent readers blinded to the clinical data. Based on the post-hoc analysis of a 6-months open-label randomized-controlled trial conducted by us (26), intra-observer reproducibility was 0.987, 0.994, 0.982, and 0.983 for erosion width, depth, volume and quantitative osteosclerosis, respectively. Inter-observer reproducibility as determined by intraclass correlation coefficient was: 0.977, 0.979, 0.962, and 0.974 for erosion width, depth, volume and quantitative osteosclerosis, respectively. Inter-reader agreement for the assessment of detecting the presence or the grade of osteosclerosis was also high (Kappa: 0.81~0.91).

# **Joint Space Width analysis**

Volumetric joint space will be quantified using an algorithm developed by consensus from the Study grouP for eXtreme Computed Tomography in Rheumatoid Arthritis (SPECTRA) [33]. The 3-D JSW including mean (JSW.Mean, mm), maximum (JSW.Max, mm), minimum (JSW.Min, mm), SD (JSW.SD, mm), asymmetry [defined as JSW.Asymm = ratio of JSW.Max/JSW.Min,] as well as volume (JSV, mm³) will be calculated. Cuts through the sagittal and coronal planes (2-dimensional) will be automatically generated for visualization. A rheumatologist with HR-pQCT expertise will review all joints and score for degree of luxation (none, subluxation, luxation) and bone-on-bone contact (yes, no).

# Ultrasound assessment of synovitis, dactylitis, enthesitis and digital pulleys

Each patient will undergo musculoskeletal ultrasound assessment of synovitis, dactylitis, enthesitis and the digital pulleys. The following anatomical sites and structures will be examined: (1) bilateral wrists, (2) bilateral metacarpophalangeal (MCP) joints 1-5, (3) bilateral proximal interphalangeal (PIP) joint 2-4, (4) interphalangeal joint of the thumbs, (4) bilateral distal interphalangeal (DIP) joints 2-4, (5) digits suspected of dactylitis, (6) digital pulleys A1, A2, A3, A4 and A5 of digits 2-4 of the more severely affected or the dominant hand if both hands are equally affected, (7) entheses including common extensor tendon at lateral epicondyle of humerus, the common flexor tendon at medial epicondyle of humerus, triceps tendon at olecranon process of ulnar, quadriceps femoris tendon at superior border of patella, patellar tendon at inferior border of patella and tibial tuberosity, Achilles tendon at calcaneus and plantar fascia at medial tubercle of calcaneus at baseline, week 24 and week 48 of follow-up. Baseline US will be performed on the same day, or within 1 week of clinical and laboratory assessment.

The US examination of each patient will be performed by 1 rheumatologist trained in musculoskeletal US and blinded to clinical and laboratory data. Each patient will undergo bilateral dynamic B-mode and power Doppler US examination.

OMERACT definitions for ultrasonographic pathologies, elementary lesions, definitions and scoring for enthesitis in spondyloarthritis and psoriatic arthritis are used (27-29). For the assessment of dactylitis, a variety of elementary lesions including flexor tendon tenosynovitis, joint synovitis, extratendinous soft tissue thickening, extensor tendonitis, enthesitis (finger extensor tendon, collateral ligaments, flexor fibrous sheaths, flexor pulleys, functional entheses), tenosynovitis, paratendonitis, synovitis, subcutaneous/peritendon tissue inflammation, proliferative and erosive bone changes will be assessed. Two measurements (transverse and longitudinal) will be done for assessing the thickness of the pulleys. The thickness of the A1, A3 and A5 pulley will be measured at the level of MCP, PIP and DIP level respectively. The A2 and A4 pulleys' thickness will be assessed in full extension, in correspondence to the proximal and middle phalanx, from their thickest sites. The US machine used is Esaote MyLab™Class-C equipped with a 6-18 MHz linear array transducer and 6-18 MHz hockey stick probe. The scanning technique will follow the European League Against Rheumatism (EULAR) standardized procedures for US imaging in rheumatology. The B-mode and power Doppler settings will be optimized and fixed for all the examinations.

# Erosion and joint space narrowing assessment by radiographs

Radiographs at baseline, 24 and 48 weeks will be obtained and assessed by one radiologist and one rheumatologist who are masked to treatment groups. Radiological progression will be assessed using the Sharp-van der Heijde modified scoring method for PsA [34]. This method is based on the Sharp-van der Heijde method for assessing erosions and joint space narrowing of joints of hands and feet in RA. In addition to the joints evaluated for rheumatoid arthritis, the distal interphalangeal joints (DIPs) of the hands are assessed. It evaluates erosions in 20 joints in each hand and wrist, and six joints in each foot. These erosions are scored on a scale of 1–5 in the hands depending on the surface area affected and 0–10 in the feet. Total erosion scores range from 0 to 200 in the hands and 0 to 120 in the feet. Joint Space Narrowing (JSN) is assessed in 20 joints in each hand and wrist, and six joints in each foot on a scale of 1–4. The score of JSN ranges from 0 to 160 in the hands and from 0 to 48 in the feet.

<u>Data processing and analysis</u> Statistical analyses will be performed using the Statistics Package for Social Sciences (SPSS). Data will be analysed in an intention-to-treat manner. Patients who discontinued treatment or violated treatment protocol will be excluded from analysis. Missing data are assumed missing at random and will be treated using a multiple Imputation method (30). Based on the pilot study and our previous experience, the missing data is estimated to be less than 5%. Descriptive statistics will be used for demographic and clinical variables included frequencies, means and standard deviations, median and interquartile range. T-test, Mann-Whitney U test and Chi-square test will be

used to evaluate differences in baseline characteristics between secukinumab group and placebo group. Changes of the outcome measurements between groups will be tested using t-test, Mann-Whitney U test, repeated measures analysis of variance (ANOVA) or Chi-square test where appropriate. Multivariate linear or logistic regression will be used to explore the association between the use of secukinumab and outcome measurements adjusting for baseline characteristics. A 2-tailed probability value of p < 0.05 is considered statistically significant.

#### Reference

- 1. Mortezavi M, Thiele R, Ritchlin C. The joint in psoriatic arthritis. Clinical and experimental rheumatology. 2015;33(5 Suppl 93):S20-5.
- 2. Kane D, Stafford L, Bresnihan B, FitzGerald O. A prospective, clinical and radiological study of early psoriatic arthritis: an early synovitis clinic experience. Rheumatology (Oxford, England). 2003;42(12):1460-8.
- 3. Acosta Felquer ML, FitzGerald O. Peripheral joint involvement in psoriatic arthritis patients. Clinical and experimental rheumatology. 2015;33(5 Suppl 93):S26-30.
- 4. Gossec L, Smolen JS, Ramiro S, de Wit M, Cutolo M, Dougados M, et al. European League Against Rheumatism (EULAR) recommendations for the management of psoriatic arthritis with pharmacological therapies: 2015 update. Annals of the rheumatic diseases. 2016;75(3):499-510.
- 5. Poggenborg RP, Bird P, Boonen A, Wiell C, Pedersen SJ, Sorensen IJ, et al. Pattern of bone erosion and bone proliferation in psoriatic arthritis hands: a high-resolution computed tomography and radiography follow-up study during adalimumab therapy. Scandinavian journal of rheumatology. 2014;43(3):202-8.
- 6. Fouque-Aubert A, Boutroy S, Marotte H, Vilayphiou N, Bacchetta J, Miossec P, et al. Assessment of hand bone loss in rheumatoid arthritis by high-resolution peripheral quantitative CT. Annals of the rheumatic diseases. 2010;69(9):1671-6.
- 7. Lee CH, Srikhum W, Burghardt AJ, Virayavanich W, Imboden JB, Link TM, et al. Correlation of structural abnormalities of the wrist and metacarpophalangeal joints evaluated by high-resolution peripheral quantitative computed tomography, 3 Tesla magnetic resonance imaging and conventional radiographs in rheumatoid arthritis. International journal of rheumatic diseases. 2015;18(6):628-39.
- 8. Finzel S, Rech J, Schmidt S, Engelke K, Englbrecht M, Schett G. Interleukin-6 receptor blockade induces limited repair of bone erosions in rheumatoid arthritis: a micro CT study. Annals of the rheumatic diseases. 2013;72(3):396-400.
- 9. Finzel S, Rech J, Schmidt S, Engelke K, Englbrecht M, Stach C, et al. Repair of bone erosions in rheumatoid arthritis treated with tumour necrosis factor inhibitors is based on bone apposition at the base of the erosion. Annals of the rheumatic diseases. 2011;70(9):1587-93.
- 10. Miossec P, Korn T, Kuchroo VK. Interleukin-17 and type 17 helper T cells. The New

England journal of medicine. 2009;361(9):888-98.

- 11. Menon B, Gullick NJ, Walter GJ, Rajasekhar M, Garrood T, Evans HG, et al. Interleukin-17+CD8+ T cells are enriched in the joints of patients with psoriatic arthritis and correlate with disease activity and joint damage progression. Arthritis & rheumatology (Hoboken, NJ). 2014;66(5):1272-81.
- 12. Mease PJ, McInnes IB, Kirkham B, Kavanaugh A, Rahman P, van der Heijde D, et al. Secukinumab Inhibition of Interleukin-17A in Patients with Psoriatic Arthritis. The New England journal of medicine. 2015;373(14):1329-39.
- 13. Finzel S, Englbrecht M, Engelke K, Stach C, Schett G. A comparative study of periarticular bone lesions in rheumatoid arthritis and psoriatic arthritis. Annals of the rheumatic diseases. 2011;70(1):122-7.
- 14. van der Heijde D, Salonen D, Weissman BN, Landewe R, Maksymowych WP, Kupper H, et al. Assessment of radiographic progression in the spines of patients with ankylosing spondylitis treated with adalimumab for up to 2 years. Arthritis research & therapy. 2009;11(4):R127.
- 15. van der Heijde D, Landewe R, Baraliakos X, Houben H, van Tubergen A, Williamson P, et al. Radiographic findings following two years of infliximab therapy in patients with ankylosing spondylitis. Arthritis and rheumatism. 2008;58(10):3063-70.
- 16. van der Heijde D, Landewe R, Einstein S, Ory P, Vosse D, Ni L, et al. Radiographic progression of ankylosing spondylitis after up to two years of treatment with etanercept. Arthritis and rheumatism. 2008;58(5):1324-31.
- 17. Finzel S, Kraus S, Schmidt S, Hueber A, Rech J, Engelke K, et al. Bone anabolic changes progress in psoriatic arthritis patients despite treatment with methotrexate or tumour necrosis factor inhibitors. Annals of the rheumatic diseases. 2013;72(7):1176-81.
- 18. Baeten D, Sieper J, Braun J, Baraliakos X, Dougados M, Emery P, et al. Secukinumab, an Interleukin-17A Inhibitor, in Ankylosing Spondylitis. The New England journal of medicine. 2015;373(26):2534-48.
- 19. Sherlock JP, Joyce-Shaikh B, Turner SP, Chao CC, Sathe M, Grein J, et al. IL-23 induces spondyloarthropathy by acting on ROR-gammat+ CD3+CD4-CD8- entheseal resident T cells. Nature medicine. 2012;18(7):1069-76.
- 20. Ono T, Okamoto K, Nakashima T, Nitta T, Hori S, Iwakura Y, et al. IL-17-producing gammadelta T cells enhance bone regeneration. Nature communications. 2016;7:10928.
- 21. Mumtaz A, Gallagher P, Kirby B, Waxman R, Coates LC, Veale JD, et al. Development of a preliminary composite disease activity index in psoriatic arthritis. Ann Rheum Dis. 2011;70(2):272-7.
- 22. Finzel S, Ohrndorf S, Englbrecht M, Stach C, Messerschmidt J, Schett G, et al. A detailed comparative study of high-resolution ultrasound and micro-computed tomography for detection of arthritic bone erosions. Arthritis and rheumatism. 2011;63(5):1231-6.

- 23. Regensburger A, Rech J, Englbrecht M, Finzel S, Kraus S, Hecht K, et al. A comparative analysis of magnetic resonance imaging and high-resolution peripheral quantitative computed tomography of the hand for the detection of erosion repair in rheumatoid arthritis. Rheumatology (Oxford, England). 2015;54(9):1573-81.
- 24. Pakdel A, Robert N, Fialkov J, Maloul A, Whyne C. Generalized method for computation of true thickness and x-ray intensity information in highly blurred sub-millimeter bone features in clinical CT images. Physics in medicine and biology. 2012;57(23):8099-116.
- 25. Bruynesteyn K, Boers M, Kostense P, van der Linden S, van der Heijde D. Deciding on progression of joint damage in paired films of individual patients: smallest detectable difference or change. Annals of the rheumatic diseases. 2005;64(2):179-82.
- 26. Wong P, Zhu TY, Qin L, Li EK, Tam L-S. AB0384 Comparison of the Effect of Denosumab and Alendronate on Bone Density and Microarchitecture at the 2ND Metacarpal Head in Rheumatoid Arthritis Females with Low Bone Mass by High- Resolution Peripheral Quantitative Computer Tomography: A Randomized Controlled Pilot Trial. Annals of the rheumatic diseases. 2015;74(Suppl 2):1021.
- 27. Wakefield RJ, Balint PV, Szkudlarek M, Filippucci E, Backhaus M, D'Agostino MA, et al. Musculoskeletal ultrasound including definitions for ultrasonographic pathology. J Rheumatol. 2005;32(12):2485-7.
- 28. Bruyn GA, Iagnocco A, Naredo E, Balint PV, Gutierrez M, Hammer HB, et al. OMERACT Definitions for Ultrasonographic Pathologies and Elementary Lesions of Rheumatic Disorders 15 Years On. J Rheumatol. 2019;46(10):1388-93.
- 29. Balint PV, Terslev L, Aegerter P, Bruyn GAW, Chary-Valckenaere I, Gandjbakhch F, et al. Reliability of a consensus-based ultrasound definition and scoring for enthesitis in spondyloarthritis and psoriatic arthritis: an OMERACT US initiative. Ann Rheum Dis. 2018;77(12):1730-5.
- 30. Rubin DB. Inference and missing data. Biometrika. 1976;63(3):581-92.

**Table 1.** The minimal disease activity (MDA) criteria of Coates, *et al (1)*. Patients are deemed to be in MDA when they meet 5 of 7 of the criteria.

| Feature | Cutoff |
|---------------------------------------|--------|
| 2 | |
| Pain by VAS, 0–100 | ≤15 |
| Global disease by VAS, 0–100 | ≤20 |
| HAQ, 0-3 | ≤0.5 |
| Tender joint count | ≤1 |
| Swollen joint count | ≤1 |
| PASI, 0-72 | ≤1 |
| OR body surface area involved, 0–100% | ≤3 |
| Enthesitis | ≤1 |

VAS: visual analog scale; HAQ: Health Assessment Questionnaire (2); PASI: Psoriasis Area and Severity Index (3). Enthesial sites assessed include the bilateral first costochondral joints, seventh costochondral joints, posterior superior iliac spines, anterior superior iliac spines, iliac crests, proximal insertion of Achilles tendons, and the fifth lumbar spinous process.

#### References:

- 1. Coates LC, Fransen J, Helliwell PS. Defining minimal disease activity in psoriatic arthritis: a proposed objective target for treatment. Ann Rheum Dis. 2010;69(1):48-53.
- Pincus T, Swearingen C, Wolfe F. Toward a multidimensional Health Assessment Questionnaire (MDHAQ): assessment of advanced activities of daily living and psychological status in the patient-friendly health assessment questionnaire format. Arthritis & Rheumatism. 1999;42(10):2220-30.
- 3. Fredriksson T, Pettersson U. Severe psoriasis--oral therapy with a new retinoid. Dermatologica. 1978;157(4):238-44



<sup>\*</sup>Treatment adjustment is allowed after week 12

<sup>#</sup> Radiological assessment include X-ray and HRpQCT

Figure 2. Quantification of the erosion volume .



c. Define the ROI including the erosion (V1) or excluding it (V2) and 3D reconstruction of the erosion.

Verosion= V1-V2; V =sum(A\_i\*0.082), where A1\_i or A2\_i is the area on slice i (mm²), including or excluding erosion, and 0.082 mm is the thickness of slice.

Figure 3. Osteosclerosis.



Typical images showing an erosion without osteosclerosis (Grade 0) at baseline, Grade 1 and Grade 2 osteosclerosis at 3 and 6 months in a pilot study, respectively.